CLINICAL TRIAL: NCT02246725
Title: Observational Study of Early Contact With Palliative Care Unit for Patients Receiving First Line Palliative Chemotherapy With Cancer in Upper Gastrointestinal Canal, or Second Line Palliative Chemotherapy in Patients With Colorectal Cancer - an Open, Randomised Investigator Initiated Trial.
Acronym: ALLAN
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MS01
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Tumor in Upper Gastrointestinal Canal or Patients With Colorectal Cancer
Keywords: Colorectal Neoplasms; Depression; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Palliative chemotherapy; Palliative care; Palliative treatment; Quality of life; Quality of life for relatives; Survival
MeSH Terms: conditions — Colorectal Neoplasms; Depression; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Contact with palliative care unit versus contact when needed.
  Interventions: Other: Contact with palliative care unit.

INTERVENTIONS:
Other: Contact with palliative care unit.

SUMMARY:
In this trial, patients with cancer in the upper gastrointestinal canal who are going to receive first line palliative chemotherapy and patients with colorectal cancer who are going to receive second line palliative chemotherapy will be included. Participating patients will be randomized between early contact with a palliative care unit, or contact with a palliative care unit when needed. The objectives with the trial is to investigate if an early establishment with a palliative care unit will have a positive impact on the patients quality of life, this also applies for the nearest relative, survival, and if a difference in numbers of chemotherapy cycles can be detected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumor in upper gastrointestinal canal, who is going to start treatment with first line palliative chemotherapy
* Patients with colorectal cancer, who is going to start treatment with second line palliative chemotherapy
* Signed written informed concent

Exclusion Criteria:

* Patients with neuroendocrine tumor
* Patients with already ongoing chemotherapy
* Patients with already established contact with palliative care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tumor in esophagus, stomach, pancreas liver-biliary passage receiving first line palliative chemotherapy, or patients with colorectal cancer receiving second line palliative chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-10; Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life, such as pain, anxiety. | At baseline, every 6th week until death (approximately 1 year). The patients relative will be followed similarly until patients death and then every 12th week for 1 year.
  Evaluation will be performed by different quality of life forms sent to the patient every 6th week, and by telephone contact with a study nurse every 6th week until patients death. The same also applies for the patients nearest relative; quality of life forms will be sent every 12th week for additional 1 year.

SECONDARY OUTCOMES:
Survival | Approximately 12 months.

OTHER OUTCOMES:
Numbers of chemotherapy cycles | Approximately 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Segerlantz, MD, PhD, Principal Investigator — Palliative Care and Advanced Home Health Care, Primary Health Care Skåne, Sankt lars väg 81, SE-221 85 LUND, Sweden
Locations (1):
- Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Bojesson A, Brun E, Eberhard J, Segerlantz M. Quality of life for patients with advanced gastrointestinal cancer randomised to early specialised home-based palliative care: the ALLAN trial. Br J Cancer. 2024 Sep;131(4):729-736. doi: 10.1038/s41416-024-02764-x. Epub 2024 Jul 1. PMID 38951699